CLINICAL TRIAL: NCT01177228
Title: A Phase 2, Randomized, Placebo-Controlled, Double-Blind Study to Determine the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of MLN0002 Following Multiple Intravenous Doses in Patients With Ulcerative Colitis
Brief Title: Study of Vedolizumab Following Multiple Intravenous Doses in Patients With Ulcerative Colitis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Millennium Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: C13002; U1111-1156-8540 (Registry Identifier: WHO)
Record Dates: First submitted 2010-08-05; First posted 2010-08-06 (Estimated); Results first posted 2014-07-18 (Estimated); Last update posted 2014-07-18 (Estimated); Status verified 2014-06

CONDITIONS: Ulcerative Colitis
MeSH Terms: conditions — Colitis, Ulcerative | interventions — vedolizumab; LDP-02

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- Placebo (Placebo Comparator): Vedolizumab-matching placebo, intravenous (IV), infusion on Days 1, 15, 29 and 85.
  Interventions: Drug: Placebo
- Vedolizumab 2 mg/kg (Experimental): Vedolizumab, 2 mg/kg, IV infusion on Days 1, 15, 29 and 85.
  Interventions: Drug: Vedolizumab
- Vedolizumab 6 mg/kg (Experimental): Vedolizumab 6 mg/kg, IV infusion on Days 1, 15, 29 and 85.
  Interventions: Drug: Vedolizumab
- Vedolizumab 10 mg/kg (Experimental): Vedolizumab 10 mg/kg, IV infusion on Days 1, 15, 29 and 85.
  Interventions: Drug: Vedolizumab

INTERVENTIONS:
Drug: Vedolizumab — Vedolizumab for intravenous infusion
  Other Names: Entyvio; MLN0002; MLN02; LDP-02
  Arms: Vedolizumab 10 mg/kg; Vedolizumab 2 mg/kg; Vedolizumab 6 mg/kg
Drug: Placebo — Placebo intravenous infusion
  Arms: Placebo

SUMMARY:
The main objectives of this study were to evaluate the safety, tolerability, pharmacokinetics (PK), and pharmacodynamics (PD) of multiple doses of vedolizumab in patients with ulcerative colitis (UC).

DETAILED DESCRIPTION:
At the end of the study, eligible participants could enroll and receive treatment and follow-up in Study C13004 (NCT00619489). Participants who did not proceed into Study C13004 were followed by telephone contact at 6-month intervals for 2 years after the last administration of study treatment to collect reports of adverse events, including colectomy, severe infections [including progressive multifocal leukoencephalopathy (PML)], and dysplasia/cancer.

ELIGIBILITY:
Inclusion Criteria:

Each patient must meet all of the following inclusion criteria to be enrolled in the study.

* Males or non-pregnant, non-lactating females voluntarily able to give informed consent
* All patients must agree to use 2 effective forms of contraception from screening to the end of the study
* Negative surveillance colonoscopy within the last 6 months if indicated by standard clinical practice guidelines
* Confirmed and active ulcerative colitis (UC)

  * Partial Mayo Score 1 - 7
  * Disease involvement extending proximal to the rectum
* May be receiving a therapeutic dose of conventional therapies for UC as defined by the protocol

Exclusion Criteria:

Patients meeting any of the following exclusion criteria are not to be enrolled in the study.

* Patients who require ulcerative colitis (UC) surgical intervention or for whom surgical intervention is anticipated during the study
* Patients who fail to meet laboratory values as specified in the protocol or have a positive progressive multifocal leukoencephalopathy (PML) subjective symptom checklist during the screening period
* Low-grade dysplasia, high-grade dysplasia, dysplasia-associated lesion or mass, or colorectal cancer
* Treatment with cyclosporine, FK506 (tacrolimus) or infliximab within 60 days prior to study
* Patients receiving any of the following within 14-days prior to the study: antibiotics for treatment of irritable bowel syndrome, heparin or warfarin, narcotics, tube feeding, defined formula diets or parenteral alimentation
* Colostomy, fistulae or known fixed symptomatic stenosis of the intestine
* Immunologic or ischemic intestinal condition
* Toxic megacolon
* Chronic hepatitis B or C or human immunodeficiency virus (HIV) infection
* Any vaccinations within 30 days prior to study drug administration
* History of imaging abnormalities, multiple sclerosis (MS), brain tumor or neurodegenerative disease
* Significantly impaired liver or renal function
* Current or recent history of alcohol dependence
* Current use of illicit drugs
* Active or recent serious infections or serious underlying disease as specified in protocol
* Active psychiatric problems that might interfere with compliance to study
* Previous exposure to MLN0002
* Participated in an investigational study within 30 days prior to study drug administration or received treatment with an investigational monoclonal antibody within the last 6 months

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 47 (Actual)
Dates: Start 2007-05; Primary Completion 2008-06 (Actual); Study Completion 2008-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Millennium Pharmaceuticals, Inc.

REFERENCES:
- [Derived] Colombel JF, Sands BE, Rutgeerts P, Sandborn W, Danese S, D'Haens G, Panaccione R, Loftus EV Jr, Sankoh S, Fox I, Parikh A, Milch C, Abhyankar B, Feagan BG. The safety of vedolizumab for ulcerative colitis and Crohn's disease. Gut. 2017 May;66(5):839-851. doi: 10.1136/gutjnl-2015-311079. Epub 2016 Feb 18. PMID 26893500
- [Derived] Rosario M, Dirks NL, Gastonguay MR, Fasanmade AA, Wyant T, Parikh A, Sandborn WJ, Feagan BG, Reinisch W, Fox I. Population pharmacokinetics-pharmacodynamics of vedolizumab in patients with ulcerative colitis and Crohn's disease. Aliment Pharmacol Ther. 2015 Jul;42(2):188-202. doi: 10.1111/apt.13243. Epub 2015 May 20. PMID 25996351

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in the study at 2 study centers in Canada and 9 study centers in Russia, from 02 May 2007 to 16 June 2008.
Pre-assignment Details: Participants with active ulcerative colitis were randomized in a 4:1 ratio of vedolizumab to placebo.
Groups:
- Placebo: Vedolizumab-matching placebo, intravenous (IV) infusion on Days 1, 15, 29 and 85.
- Vedolizumab 2 mg/kg: Vedolizumab 2 mg/kg, IV infusion on Days 1, 15, 29 and 85.
- Vedolizumab 6 mg/kg: Vedolizumab 6 mg/kg IV infusion on Days 1, 15, 29 and 85.
Period: Overall Study
Arm/Group | Placebo | Vedolizumab 2 mg/kg | Vedolizumab 6 mg/kg | Vedolizumab 10 mg/kg
Started | 9 | 13 | 14 | 11
Received Treatment | 9 | 12 | 14 | 11
Completed | 8 | 11 | 14 | 11
Not Completed | 1 | 2 | 0 | 0
Not completed — Positive tuberculosis test | 0 | 1 | 0 | 0
Not completed — Worsening disease activity | 1 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Baseline measures are reported for the Safety Analysis Set - all enrolled participants who received at least 1 dose of study treatment. One participant was randomized but not dosed and is not included in this population.
Groups:
- Placebo: Vedolizumab-matching placebo, intravenous (IV), one 30-minute infusion on Days 1, 15, 29 and 85.
- Vedolizumab 2 mg/kg: Vedolizumab 2 mg/kg IV infusion on Days 1, 15, 29 and 85.
- Vedolizumab 10 mg/kg: Vedolizumab 10 mg/kg IV infusion on Days 1, 15, 29 and 85.
- Total: Total of all reporting groups
Arm/Group | Placebo | Vedolizumab 2 mg/kg | Vedolizumab 6 mg/kg | Vedolizumab 10 mg/kg | Total
Number analyzed (Participants) | 9 | 12 | 14 | 11 | 46
Age, Continuous [Mean (Standard Deviation); unit: years] | 34.2 (8.11) | 39.0 (6.06) | 44.4 (12.37) | 44.3 (14.99) | 41.0 (11.46)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 8 | 7 | 6 | 27
  Male | 3 | 4 | 7 | 5 | 19
Race/Ethnicity, Customized [Number; unit: participants]
  White, Not Hispanic or Latino | 9 | 12 | 14 | 11 | 46
Height [Mean (Standard Deviation); unit: cm] | 168.0 (7.33) | 169.8 (10.52) | 167.9 (9.87) | 170.7 (8.15) | 169.1 (9.00)
Weight [Mean (Standard Deviation); unit: kg] | 74.01 (24.04) | 75.76 (20.98) | 79.61 (16.65) | 73.46 (13.60) | 76.04 (18.38)
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m²] | 26.22 (8.46) | 26.03 (5.58) | 28.51 (6.66) | 25.29 (5.07) | 26.64 (6.37)
Body Surface Area (BSA) [Mean (Standard Deviation); unit: m²] | 1.84 (0.31) | 1.88 (0.30) | 1.92 (0.21) | 1.86 (0.20) | 1.88 (0.25)
Time Since Onset of Symptoms [Mean (Standard Deviation); unit: years] | 3.92 (2.79) | 6.25 (5.00) | 6.85 (4.31) | 7.03 (10.13) | 6.16 (6.08)
Time Since Diagnosis [Mean (Standard Deviation); unit: years] | 2.29 (2.43) | 5.26 (4.92) | 5.38 (4.79) | 5.46 (9.72) | 4.76 (6.01)
Participants with Acute Exacerbations in Past 12 Months [Number; unit: participants]
  Yes | 9 | 12 | 13 | 9 | 43
  No | 0 | 0 | 1 | 2 | 3
Participants Hospitalized for UC in Past 12 Months [Number; unit: participants]
  Yes | 5 | 3 | 2 | 4 | 14
  No | 4 | 9 | 12 | 7 | 32
Participants with Ongoing Therapy for UC at Enrollment [Number; unit: participants]
  Yes | 9 | 11 | 13 | 9 | 42
  No | 0 | 1 | 1 | 2 | 4
Participants with Significant Medical Conditions in Past 6 Months [Number; unit: participants]
  Yes | 5 | 11 | 12 | 9 | 37
  No | 4 | 1 | 2 | 2 | 9

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Adverse Events
Description: An adverse event (AE) is any untoward medical occurrence in a patient administered a pharmaceutical product, which does not necessarily have a causal relationship with the treatment. The investigator systematically collected information adequate to determine both the outcome and severity of the AE, and whether or not it was drug-related or met the criteria for classification as a serious adverse event (SAE). An SAE was defined as an AE that resulted in (or posed risk for) death, inpatient hospitalization (or prolonging hospitalization), or congenital, persistent or significant disability/incapacity.
  The intensity for each AE was defined according to the following criteria:
  Mild: Awareness of sign or symptom, but easily tolerated Moderate: Discomfort enough to cause interference with normal daily activities Severe: Inability to perform normal daily activities.
Time Frame: From the first date of study drug administration through Day 253
Population: Safety Analysis Set, defined as all enrolled participants who received at least 1 dose of study treatment. One participant was randomized but not dosed and is not included in this population.
Measure: Number; unit: participants
Arm/Group | Placebo | Vedolizumab 2 mg/kg | Vedolizumab 6 mg/kg | Vedolizumab 10 mg/kg
Number analyzed (Participants) | 9 | 12 | 14 | 11
participants
  Any Adverse Event | 7 | 9 | 9 | 6
  Severe Adverse Event | 0 | 0 | 1 | 1
  Drug-related Adverse Event | 3 | 2 | 1 | 1
  Serious Adverse Event | 0 | 1 | 0 | 1
  Drug-related Serious Adverse Event | 0 | 0 | 0 | 0
  Serious Adverse Event Resulting in Discontinuation | 0 | 0 | 0 | 0
  On-study Deaths | 0 | 0 | 0 | 0

2. Primary Outcome: Cmax: Maximum Observed Plasma Concentration of Vedolizumab on Days 1 and 85
Description: Maximum observed plasma concentration (Cmax) is the peak plasma concentration of a drug after administration, obtained directly from the plasma concentration-time curve.
Time Frame: Days 1 and 85, prior to and 2, 12, 24, 48, and 72 hours after dosing.
Population: Pharmacokinetic (PK) Analysis Set, defined as all vedolizumab participants for whom there were sufficient data to estimate PK. Analyses only include participants with available data at each time point (indicated by "n").
Measure: Mean (Standard Deviation); unit: µg/mL
Groups:
- Vedolizumab (6 mg/kg): Vedolizumab 6 mg/kg IV infusion on Days 1, 15, 29 and 85.
Arm/Group | Vedolizumab 2 mg/kg | Vedolizumab (6 mg/kg) | Vedolizumab 10 mg/kg
Number analyzed (Participants) | 10 | 14 | 11
µg/mL
  Cmax, Day 1 (n=10, 14, 11) | 54.0 (8.9) | 154.3 (41.5) | 279.0 (167.9)
  Cmax, Day 85 (n=9, 14, 11) | 60.4 (12.5) | 191.9 (42.6) | 291.9 (95.0)

3. Primary Outcome: Cmin: Minimum Observed Plasma Concentration of Vedolizumab
Description: Minimum observed plasma concentration (Cmin) is the lowest plasma concentration of a drug after administration, obtained directly from the plasma concentration-time curve.
Time Frame: Day 85, prior to and 2, 12, 24, 48, and 72 hours after dosing.
Population: PK Analysis Set; participants with available data.
Measure: Mean (Standard Deviation); unit: μg/mL
Arm/Group | Vedolizumab 2 mg/kg | Vedolizumab 6 mg/kg | Vedolizumab 10 mg/kg
Number analyzed (Participants) | 9 | 14 | 11
μg/mL | 7.25 (2.41) | 29.33 (13.36) | 44.74 (19.80)

4. Primary Outcome: Area Under the Plasma Concentration-Time Curve (AUC) for Vedolizumab
Description: AUC was calculated for 3 time intervals during the study:
  1. AUC (Day 0-14): from administration on Day 0 to last quantifiable concentration on Day 14, selected to capture the AUC following the first dose of vedolizumab until administration of the second dose
  2. AUC(Day 85-99): from administration on Day 85 to last quantifiable concentration on Day 99, selected to assess the amount of drug accumulation with the planned loading regimen by comparing it to AUC(Day 0-14)
  3. AUC(Day 85-141): from the first quantifiable concentration on Day 85 to the last quantifiable concentration on Day 141, selected to assess the drug exposure over an 8-week period
Time Frame: Days 0-14, Days 85-99, Days 85-141
Population: PK Analysis Set; participants with available data at each time point (indicated by "n").
Measure: Mean (Standard Deviation); unit: day*μg/mL
Arm/Group | Vedolizumab 2 mg/kg | Vedolizumab 6 mg/kg | Vedolizumab 10 mg/kg
Number analyzed (Participants) | 10 | 14 | 11
day*μg/mL
  AUC (Day 0-14) (n=10, 14, 11) | 375 (59) | 1058 (270) | 1765 (822)
  AUC(Day 85-99) (n=9, 14, 11) | 473 (92) | 1532 (227) | 2608 (795)
  AUC(Day 85-141) (n=9, 14, 11) | 1082 (243) | 3318 (698) | 5633 (1927)

5. Primary Outcome: Terminal Phase Elimination Half-life (t½) of Vedolizumab
Description: Terminal phase elimination half-life (t½) is the time required for half of the drug to be eliminated from the plasma.
Time Frame: Pre-dose through Day 253
Population: PK Analysis Set; participants with available data
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Vedolizumab 2 mg/kg | Vedolizumab 6 mg/kg | Vedolizumab 10 mg/kg
Number analyzed (Participants) | 9 | 14 | 11
days | 15.1 (2.0) | 22.0 (6.7) | 20.6 (7.2)

6. Primary Outcome: Maximum Drug Effect (Emax) of Vedolizumab as Measured by Percent Inhibition of the Act-1 Marker
Description: The target of vedolizumab is α4β7 integrin, a receptor found on inflammatory immune cells that guides these inflammatory cells to the gut and binds to the Mucosal Addressin Cell Adhesion Molecule-1 (MAdCAM-1) on gut endothelial cells. The extent of the α4β7 receptor saturation by vedolizumab was assessed using the Act-1 binding interference assay. Act-1 is a mouse antibody similar to vedolizumab that also binds α4β7 integrin. The assay measures the percent inhibition of the Act-1 due to the presence of vedolizumab binding.
  Emax was calculated on Day 1, Day 85 and based on all available data.
Time Frame: Days 1, 2, 3, 4, 8, 15, 29, 43, 57, 71, 85, 86, 87, 89, 92, 99, 113, 127, 141, 155, 169, 183, 197, 211, 225, 239, and 253
Population: Pharmacodynamic (PD) Analysis Set, defined as all participants for whom there were sufficient data to estimate PD. Analyses only include participants with available data (indicated by "n").
Measure: Mean (Standard Deviation); unit: percent inhibition
Groups:
- Placebo: Vedolizumab-matching placebo IV infusion on Days 1, 15, 29 and 85.
Arm/Group | Placebo | Vedolizumab 2 mg/kg | Vedolizumab 6 mg/kg | Vedolizumab 10 mg/kg
Number analyzed (Participants) | 8 | 10 | 12 | 11
percent inhibition
  Day 1 (n=8, 10, 12, 11) | 18.4 (19.3) | 98.0 (1.1) | 99.0 (0.8) | 98.3 (1.3)
  Day 85 (n=8, 9, 12, 11) | 22.8 (15.3) | 98.7 (1.2) | 99.1 (0.7) | 98.6 (0.8)
  All available (n=8, 10, 12, 11) | 56.3 (29.4) | 99.5 (0.6) | 99.8 (0.3) | 99.8 (0.3)

7. Primary Outcome: Maximum Drug Effect (Emax) as Measured by Inhibition of the MAdCAM-1-Fc Marker
Description: The target of vedolizumab is α4β7 integrin, a receptor found on inflammatory immune cells that guides these inflammatory cells to the gut and binds to the mucosal addressin cell adhesion molecule-1 (MAdCAM-1) on gut endothelial cells. The extent of the α4β7 receptor saturation by vedolizumab was assessed using the MAdCAM-1-Fc binding interference assay. MAdCAM-1-Fc is a fusion of human MAdCAM-1 with parts of a mouse monoclonal antibody. The assay measures the percent inhibition of the MAdCAM-1-Fc binding to α4β7 integrin due to the presence of vedolizumab binding.
  Emax was calculated on Day 1, Day 85, and based on all available data.
Time Frame: as for outcome 6
Population: PD Analysis Set; participants with available data (indicated by "n")
Measure: Mean (Standard Deviation); unit: percent inhibition
Arm/Group | Placebo | Vedolizumab 2 mg/kg | Vedolizumab 6 mg/kg | Vedolizumab 10 mg/kg
Number analyzed (Participants) | 8 | 10 | 11 | 10
percent inhibition
  Day 1 (n=8, 10, 11, 10) | 11.9 (15.3) | 96.4 (1.8) | 89.8 (29.8) | 96.8 (2.9)
  Day 85 (n=8, 9, 11, 10) | 8.5 (7.9) | 98.3 (1.1) | 98.3 (2.3) | 96.2 (2.6)
  All available (n=8, 10, 11, 10) | 43.3 (27.3) | 99.3 (0.6) | 99.8 (0.3) | 99.3 (0.7)

8. Primary Outcome: Area Under the Drug Effect Time Curve [AUEC(0-last)] as Measured by Inhibition of the ACT-1 Marker
Description: AUEC (0-last) is the area under the drug effect-time curve until the last available time point. Mean percent inhibition over time [AUEC(0-last)] was determined for the Act-1 marker. Act-1 is a mouse antibody similar to vedolizumab that also binds α4β7 integrin.
Time Frame: as for outcome 6
Population: PD Analysis Set; participants with available data (indicated by "n")
Measure: Mean (Standard Deviation); unit: percent inhibition*days
Arm/Group | Placebo | Vedolizumab 2 mg/kg | Vedolizumab 6 mg/kg | Vedolizumab 10 mg/kg
Number analyzed (Participants) | 8 | 10 | 12 | 11
percent inhibition*days | 4281.7 (3035.3) | 20195.9 (3814.2) | 22675.2 (2211.8) | 23613.7 (1574.4)

9. Primary Outcome: Area Under the Drug Effect Time Curve [AUEC(0-last)] as Measured by Inhibition of the MAdCAM-1-Fc Marker
Description: AUEC (0-last) is the area under the drug effect-time curve until the last available time point. Mean percent inhibition over time [AUEC(0-last)] was determined for the MAdCAM-1-Fc marker. MAdCAM-1-Fc is a fusion of human MAdCAM-1 with parts of a mouse monoclonal antibody.
Time Frame: as for outcome 6
Population: PD Analysis Set; participants with available data (indicated by "n")
Measure: Mean (Standard Deviation); unit: percent inhibition*days
Arm/Group | Placebo | Vedolizumab 2 mg/kg | Vedolizumab 6 mg/kg | Vedolizumab 10 mg/kg
Number analyzed (Participants) | 8 | 10 | 11 | 10
percent inhibition*days | 2139.2 (1513.4) | 18802.0 (3556.1) | 22322.1 (1974.2) | 22484.6 (1716.0)

ADVERSE EVENTS:
Time Frame: Adverse events were collected through Day 253 or the final study visit.
Arm/Group | Placebo | Vedolizumab 2 mg/kg | Vedolizumab 6 mg/kg | Vedolizumab 10 mg/kg
Serious Adverse Events (participants affected / at risk) | 0/9 | 1/12 | 0/14 | 1/11
Other Adverse Events (participants affected / at risk) | 7/9 | 9/12 | 9/14 | 6/11
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=9) | Vedolizumab 2 mg/kg (N=12) | Vedolizumab 6 mg/kg (N=14) | Vedolizumab 10 mg/kg (N=11)
Gastroduodenitis (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Spinal compression fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=9) | Vedolizumab 2 mg/kg (N=12) | Vedolizumab 6 mg/kg (N=14) | Vedolizumab 10 mg/kg (N=11)
Upper respiratory tract infection (Infections and infestations) | 3 | 1 | 1 | 1
Nasopharyngitis (Infections and infestations) | 1 | 2 | 1 | 0
Gastroenteritis (Infections and infestations) | 0 | 0 | 0 | 1
Infectious mononucleosis (Infections and infestations) | 0 | 0 | 1 | 0
Laryngotracheitis (Infections and infestations) | 0 | 0 | 0 | 1
Pharyngitis streptococcal (Infections and infestations) | 0 | 0 | 1 | 0
Pyelonephritis chronic (Infections and infestations) | 0 | 0 | 0 | 1
Respiratory tract infection viral (Infections and infestations) | 0 | 1 | 0 | 0
Sinusitis (Infections and infestations) | 0 | 1 | 0 | 0
Herpes zoster (Infections and infestations) | 1 | 0 | 0 | 0
Lobar pneumonia (Infections and infestations) | 1 | 0 | 0 | 0
Mastitis (Infections and infestations) | 1 | 0 | 0 | 0
Respiratory tract infection (Infections and infestations) | 1 | 0 | 0 | 0
Colitis ulcerative (Gastrointestinal disorders) | 4 | 2 | 1 | 0
Constipation (Gastrointestinal disorders) | 1 | 0 | 0 | 1
Abdominal pain upper (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Anal discomfort (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Gastritis erosive (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Gastroduodenitis (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Nausea (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Dyspepsia (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Headache (Nervous system disorders) | 1 | 2 | 3 | 2
Dizziness (Nervous system disorders) | 1 | 0 | 0 | 1
Balance disorder (Nervous system disorders) | 0 | 0 | 0 | 1
C-reactive protein increased (Investigations) | 1 | 1 | 0 | 0
Blood glucose increased (Investigations) | 0 | 0 | 1 | 0
Blood pressure increased (Investigations) | 0 | 0 | 1 | 0
Liver function test abnormal (Investigations) | 0 | 0 | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2 | 0
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1 | 0
Increased upper airway secretion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Osteoporosis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Tendonitis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Influenza like illness (General disorders) | 0 | 0 | 2 | 0
Pyrexia (General disorders) | 0 | 0 | 2 | 0
Chills (General disorders) | 0 | 0 | 1 | 0
Muscle strain (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Spinal compression fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Calculus urinary (Renal and urinary disorders) | 0 | 0 | 1 | 0
Nephrolithiasis (Renal and urinary disorders) | 0 | 0 | 0 | 1
Alopecia (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
Drug eruption (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
Hypertension (Vascular disorders) | 0 | 0 | 1 | 1
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0
Hypochromic anaemia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0
Breast adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The first study related publication will be a multi-center publication submitted within 24 months after conclusion or termination of a study at all sites. After such multi-site publication, all proposed site publications and presentations will be submitted to sponsor for review 60 days in advance of publication. Site will remove Sponsor confidential information unrelated to study results. Sponsor can delay a proposed publication for another 60 days to preserve intellectual property.